CLINICAL TRIAL: NCT02444429
Title: Evaluation of a Strategy Based on the 3-month Screening Biopsy to Optimize the Immunosuppression in Renal Transplantation: the I4BiS Study
Brief Title: 3-month Screening Biopsy to Optimize the Immunosuppression in Renal Transplantation
Acronym: I4BiS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014.848; 2014-005425-13 (EudraCT Number)
Record Dates: First submitted 2015-03-25; First posted 2015-05-14 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Renal Transplantation
Keywords: Screening renal biopsy; Immunosuppression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sub-study A experimental arm (Experimental): This experimental arm corresponds to patients with "borderline" infiltrates at 3 months, who will be randomized to receive a treatment for rejection (intensification of the corticotherapy with corticosteroid boluses = Corticosteroid boluses Methylprednisolone )
  Interventions: Drug: Corticosteroid boluses Methylprednisolone
- Sub-study A control arm (Active Comparator): This control arm corresponds to patients with "borderline" infiltrates at 3 months, who will be randomized to not change their immunosuppressive treatment (No therapeutic modification)
  Interventions: Other: No therapeutic modification
- Sub-study B experimental arm (Experimental): This experimental arm corresponds to patients without significant infiltrates 3 months, who will be randomized to stop maintenance corticotherapy (Stop maintenance corticotherapy )
  Interventions: Other: Stop maintenance corticotherapy
- Sub-study B control arm (Active Comparator): This control arm corresponds to patients without significant infiltrates 3 months, who will be randomized to not change their immunosuppressive treatment (No therapeutic modification)
  Interventions: Other: No therapeutic modification

INTERVENTIONS:
Drug: Corticosteroid boluses Methylprednisolone — Intensification of the corticotherapy in accordance with the validated protocol for the treatment of "classic" and subclinical acute rejections: 3 bolus Methylprednisolone 500 mg IV at D1, D2 and D3 then decreasing during 10-15 days at 1mg/kg/d and down to the maintenance dose.
  An anti-pneumocystis and anti-CMV prophylaxis will be systemically introduced for 3 months.
  The rest of maintenance immunosuppressive regimen (mycophenolate mofetil and anti-calcineurin) will remain unaltered
  Arms: Sub-study A experimental arm
Other: No therapeutic modification — No therapeutic modification: continuation of the corticotherapy at the maintenance dose and maintaining unaltered the rest of immunosuppressive treatment (mycophenolate mofetil and anti-calcineurin).
  Arms: Sub-study A control arm; Sub-study B control arm
Other: Stop maintenance corticotherapy — Immediate withdrawal of maintenance corticotherapy. Maintaining unaltered the rest of immunosuppressive treatment (mycophenolate mofetil and anti-calcineurin).
  Arms: Sub-study B experimental arm

SUMMARY:
Renal transplantation represents currently the best therapeutic alternative for end-stage renal failure, not only in terms of patient outcomes (better quality of life and longer survival), but also in terms of costs for the society.

Progress achieved in the last 20 years has resulted in a drastic reduction of the incidence of "classic" (i.e. clinically patent) acute cellular rejection episodes.

Unfortunately, and rather unexpectedly, this progress has had hardly any effect on the frequency of the loss of kidney transplants beyond the first year, as shown by the stagnation of grafts' half lives.

Furthermore, the use of immunosuppressant combinations that are more and more powerful has an impact on adverse effects in recipients, including an increased incidence of infections, cancers, but also metabolic complications (diabetes, osteoporosis, dyslipidemia, etc.), which are cause of significant morbi-mortality.

In an attempt to improve on these disappointing outcomes, some teams have offered to perform screening biopsies: i.e. routine biopsies at specific time points during the follow up, irrespective of graft function. Their primary interest is to allow a pathological analysis of the graft at an early stage, i.e. when potential histological lesions allow for a diagnosis but before these lesions impact on graft's function. Indeed, it has been clearly demonstrated that therapeutic adjustments intended to protect the grafts are most effective when introduced early. There is a fairly broad consensus to perform these biopsies three months and one year after the transplantation. Performing screening biopsies has led to the identification of "subclinical" forms of rejection, i.e. graft infiltration by recipient immune effectors meeting the Banff histological criteria, but without increase in creatininemia.

Assuming that about 10% of screening biopsies performed at 3 months reveal a subclinical rejection, which needs to be treated, the management strategy for the remaining 90% of patients, whose biopsies show either i) a mild inflammatory infiltrates: i.e. "borderline changes", or ii) the complete absence of immune effectors in the graft is, poorly standardized.

The investigators therefore propose to conduct a prospective randomized trial to answer these questions simultaneously by evaluating a strategy to optimize the immunosuppression of renal graft recipients based on the presence or absence of subclinical intragraft inflammatory infiltrates in the screening biopsy performed at 3 months post transplantation. Patients with borderline changes (sub-study A) will be randomized to receive a treatment for rejection (corticosteroid boluses). Patients without inflammation in their graft (sub-study B) will be randomized for corticosteroid withdrawal. Impact on graft function, progression of histological lesions and incidence of morbidity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Common to both sub-studies (A and B)

   * Renal transplant patient aged between 18 and 75.
   * Patient who received a first or second renal graft
   * Immunosuppressive treatment consisting of an anti-calcineurin [cyclosporine (trough levels: 150<T0<300)], or tacrolimus (trough levels: 8<T0<12), mycophenolate mofetil and corticosteroids.
   * Patient who benefited from a screening renal biopsy 3 months after the graft
   * Patient who gave their informed consent
   * Patient affiliated to a social security scheme or being a beneficiary of such a scheme
2. Specific to sub-study A

   * Presence of "borderline" inflammatory infiltrates on the screening biopsy at 3 months as defined by the Banff classification 2013:
   * Absence of vascular lesions (v0) and:

     * tubulitis regardless of its significance (t1-3) with minimum interstitial infiltrate (i0-i1) OR
     * interstitial infiltrates (i2-3) without significant tubulitis (≤ t1)
3. Specific to sub-study B Absence of significant inflammatory infiltrates (i0-1 and t0) on the screening biopsy at 3 months

Exclusion Criteria:

1. Common to both sub-studies (A and B)

   * Histological subclinical rejection criteria on the screening biopsy at 3 months (Banff 2009: > i2+t2)
   * Donor specific antibodies in historical serum or de novo appearance during the first 3 months
   * Humoral lesions on the 3-month biopsy (Banff score g+ptc>2)
   * "Classic" acute rejection episode proven by biopsy during the first 3 months
   * Multiorgan transplantation
   * 3rd (or subsequent) renal transplantation
   * BK virus-associated nephropathy on the screening biopsy
   * Contraindication to the 1-year screening biopsy
2. Specific to sub-study B Initial nephropathy with a high risk of recurrence on corticosteroid withdrawal: segmental and focal and segmental glomerulosclerosis, lupus nephritis, vasculitis, or membranous glomerulonephritis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Evolution of graft inflammatory lesions | 9 months
  Interstitial infiltrate (i) and tubulitis (t) will be scored at 3 months and 1 year post transplantation using Banff classification (patients will be recruted 3 months after transplantation)
  A) Patient with "borderline" infiltrates at 3 months will be randomized to receive a treatment for rejection (sub-study A), with the aim of demonstrating the superiority of this strategy in terms of infiltrates involution (superiority study).
  B) Patient without significant infiltrates at 3 months will be randomized for maintenance corticotherapy withdrawal (sub-study B), with the aim of showing that this strategy does not cause an increase in the percentage of "borderline" infiltrates compared to the strategy that maintains the corticotherapy (non-inferiority study).

SECONDARY OUTCOMES:
Graft function at 1 year post-transplantation | 9 months
  Measurement of the glomerular filtration rate by iohexol clearance at 1 year post transplantation (unit: ml/min:1.73m2)
Graft function at 1 year post-transplantation | 9 months
  Evolution of proteinuria between 3 months and 1 year (unit: g/24h).
Evolution of chronic histological lesions | 9 months
  Interstitial fibrosis will be quantified at 3 months and 1 year using a computerized color image analysis technique (unit = % fibrosis = 100*(green interstitial pixels / total interstitial pixels))
Evolution of chronic histological lesions | 9 months
  The 4 basic chronic lesions (unit = chronic glomerular damage [cg]; interstitial fibrosis [ci]; tubular fibrosis [ct]; vascular intimal thickening [cv]) will be scored at 3 months and 1 year using Banff classification)
Evaluation of the immunological risk associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Percentage of patients showing the appearance of donor specific anti-HLA antibodies using the Luminex method® between the randomization (3 months) and the end of follow-up (1 year). (unit = % of patient)
Evaluation of the immunological risk associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Proportion of patients showing an increase in humoral lesions (Banff score g+ptc) ≥ 2 on the screening biopsy at 1-year between the randomization (3 months) and the end of follow-up (1 year). (unit = % of patient)
Evaluation of the immunological risk associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Proportion of patients showing ≥ 1 acute rejection episodes (cellular or humoral) proven by biopsy between the randomization (3 months) and the end of follow-up (1 year). (unit = % of patient)
Evaluation of the metabolic tolerance profile associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Comparison of the data from the Holter monitor taken between 3 months and 1 year post-transplantation. (unit = mm of Hg)
Evaluation of the metabolic tolerance profile associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Comparison of the data from the orally induced hyperglycemia test taken between 3 months and 1 year post-transplantation. (unit = mmol/l)
Evaluation of the metabolic tolerance profile associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Comparison of the data from the lipid profile taken between 3 months and 1 year post-transplantation. (unit = mmol/l)
Evaluation of the metabolic tolerance profile associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Comparison of the data from the bone mineral density, taken between 3 months and 1 year post-transplantation. (unit = g/cm2)
Evaluation of the infectious tolerance profile associated with the different strategies of corticosteroid treatment adaptation | 9 months
  Number of infectious episodes requiring treatment during the follow-up period between the randomization (3 months) and the end of follow-up (1 year). (unit = nb of episode)
Evaluation of the impact of the different strategies for corticosteroid use on quality of life. | 9 months
  Evolution of the patients' quality of life using self-questionnaires, adapted and validated for the French language (SF36), between the randomization (3 months) and the end of follow-up (1 year). (unit = SF 36 score)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier THAUNAT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (8):
- France (8):
  - Service de Néphrologie,Transplantation, Dialyse I - Hôpital Pellegrin - CHU Bordeaux, Bordeaux
  - Service de Néphrologie, Hémodialyse, Transplantations Rénales - Hôpital de la Cavale Blanche - CHU de Brest, Brest
  - Service de Néphrologie - Hôpital Claude Huriez - CHU de Lille, Lille
  - Service de Néphrologie, Transplantation et Immunologie Clinique - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Institut de Transplantation, Urologie et Néphrologie (ITUN) - CHU de Nantes, Nantes
  - Service de Transplantation - Hôpital Universitaire Necker, Paris
  - Service de Néphrologie et Transplantation - Nouvel Hôpital Civil - CHRU Strasbourg, Strasbourg
  - Département de Néphrologie et Transplantation d'Organes - Hôpital Rangueil - CHU de Toulouse, Toulouse